CLINICAL TRIAL: NCT03986164
Title: Implants Immediately Installed in Esthetic Area With Computer-guided Surgery: Randomized Clinical Trial
Brief Title: Implants Immediately Installed in Esthetic Area With Computer-guided Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, Full professor, department of Periodontics, Piracicaba Dental School, State University of Campinas (UNICAMP), Piracicaba, São Paulo, Brazil, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09409619.3.0000.5418
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Dental Implants
Keywords: Guided Surgery; Linear Shifts; Angular Shifts; Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This is a longitudinal parallel randomized clinical trial, in Piracicaba Dental School, State University of Campinas (FOP-UNICAMP), periodic follow-ups will be performed for one year after the installation of implants in the anterior maxilla, by means of computer-assisted dental implant surgery or conventional surgery. The study will be conducted according to the Helsinki Declaration (2008), following the protocol for randomized clinical trials (Consort) (Schulz et al., 2010). The implant placement evaluations; radiographic and clinical evaluations of peri-implant tissues; as well as the success of the implants and the rehabilitation will be carried out immediately, 6 and 12 months after the implant installation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participating individuals will be allocated within each group through a computer-generated list, stored in a brown opaque envelope, under the care of an individual (TCB) other than the examiner. Only the professional responsible for the treatments will have access to the codes and both the patients and the examiners will be blind to the group to which each patient belongs, making possible the characterization of the study as double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guided surgery (GS) (Active Comparator): Installation of dental implant with the aid of the virtually planned guide by means of specific software
  Interventions: Device: Guided surgery with bovine spongious bone substitute
- Conventional surgery (CS) (Active Comparator): Installation of dental implant performed freehand using a conventional surgical guide made by study models
  Interventions: Device: Conventional surgery with bovine spongious bone substitute

INTERVENTIONS:
Device: Guided surgery with bovine spongious bone substitute — A minimally traumatic extraction will be performed aiming at the preservation of tissue integrity. After this step, milling will be performed using a sequence of guides and cutters recommended by the Raptor Implacil / Bioparts (Implacil De Bortoli) system manufacturer for implant installation (Cone Morse 3.5mm from 11-13mm Implacil De Bortoli) in computer-guided surgeries.
  In the spaces between the implant and the buccal bone plate will be filled with xenogene biomaterial (Geistlich Bio-Oss 0.25-1mm). Immediately after implant installation, the prosthetic component (Smart Line, Trunnion CM 3.5mm - T 1.5-3.5mm, height 4mm - Implacil De Bortoli) will be placed.
  If necessary, the sutures of the surgical procedures will be performed with polygalactin 5.0 (Vycril Rapid®, Jonhson's Jonhson, São José dos Campos) and will be removed after 7 days.
  Arms: Guided surgery (GS)
Device: Conventional surgery with bovine spongious bone substitute — The sequence of cutters recommended by the manufacturer for this type of surgery and installation of the same type of implant (Cone Morse due cone 3.5mm) will be adopted. The perforations of the collar for future insertion of the implants will be performed aiming the installation of the implants with its platform installed with sub-crestal position. The implant should be installed along the palatine wall to obtain primary stability, at the center of the mesio-distal width predetermined by the final restoration, with a minimum distance of 2 mm from the adjacent tooth, and 3 mm from the free gingival margin, becoming slightly palatinate (Kan et al, 2018). Immediately after installation, the prosthetic component (Smart Line, Trunnion CM 3.5mm - T 1.5-3.5mm, height 4mm) will be placed. If necessary, the sutures of the surgical procedures will be performed with polygalactin 5.0 (Vycril Rapid®, Jonhson's Jonhson, São José dos Campos) and will be removed after 7 days.
  Arms: Conventional surgery (CS)

SUMMARY:
The objective of this randomized and longitudinal clinical study is to compare the installation of immediate implants in the esthetic zone through computer-guided-surgery and conventional surgery. To this end, 22 patients who need implant-supported replacement on the anterior region of the maxilla will be selected and after extraction will receive: Guided surgery (GS): installation of dental implant with the aid of the virtually planned guide by means of specific software; Conventional surgery (CS): installation of dental implant performed freehand using a conventional surgical guide made by study models.

DETAILED DESCRIPTION:
The objective of this randomized and longitudinal clinical study is to compare the installation of immediate implants in the esthetic zone through computer-guided-surgery and conventional surgery. To this end, 22 patients who need implant-supported replacement on the anterior region of the maxilla will be selected and after extraction will receive: Guided surgery (GS): installation of dental implant with the aid of the virtually planned guide by means of specific software; Conventional surgery (CS): installation of dental implant performed freehand using a conventional surgical guide made by study models. Tomographies will be performed 10 days after the surgery for the measurement of both linear and angular shifts between the installed implants and the virtual planning. All the clinical and radiographic assessments (Plaque and Bleeding Index, Drilling Depth, Relative Clinical Insertion Level and the Margin Position of Peri-Implant Mucosa) will be carried out after the surgery and within 6 and 12 months of post-operative. Assesments of the esthetic success (pink/white score) and survival and success of the implant will also be carried out. In the prosthetic part, it will be assessed the abutment mobility; corrective measures for the prothesis; repair on prothesis or abutment. The success and survival assessments of crowns will be done through structure fracture, occlusal roughness, marginal integrity and contour of the restoration. It will also be assessed the procedural impact in quality of life by applying a 36-closed-question-survey focused on appearence, pain, oral comfort, general performance, feeding and chewing. Subsequently, the data will be tabulated, and according to their distribution, the appropriate statistical tests will be applied, considering a 5% index of significance to all the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sufficient bone volume availability apically and palatally that allows the correct positioning of the implants (Kan et al, 2011);
* Implants with primary stability of 20-45 N (Gallucci et al, 2014);
* Patients with teeth to be extracted in the Class I, II or III corono-radicular position, according to Kan et al. (2011);
* Patients with distance from the bone crest to the point of contact in adjacent teeth less than or equal to 6.5mm (Buser et al 2017).

Exclusion Criteria:

* Presence of diabetes, blood disorders and systemic diseases that prevent the surgical procedure;
* History of radiotherapy in the head or neck region;
* History of treatment with bisphosphonates;
* Pregnant or lactating women;
* Patients with teeth to be extracted in the Class V corono-radicular position, according to Kan et al. (2011);
* Gingival recession in the teeth indicated for exodontia (Kan et al, 2001);
* Acute infection at the implant site (Morton et al, 2014);
* Unavailability to attend the FOP / UNICAMP on the pre-determined days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Position of the implant | Baseline, 10 days
  Difference between angular position of the implant by computer software and angular position of the implant by free hand.

SECONDARY OUTCOMES:
Relative gingival margin position | Immediately after surgery, 6 months, 12 months
  Distance from stent probing to peri-implant margin tissue
Peri-implant probing depth | Immediately after surgery, 6 months, 12 months
  Distance from peri-implant mucosa to more apical portion of peri-implant sulcus
Relative clinical attachment level | Immediately after surgery, 6 months, 12 months
  Distance from stent probing to more apical portion of peri-implant sulcus

CONTACTS AND LOCATIONS:
Overall Officials: Enilson A Sallum, PhD, Study Chair — Piracicaba Dental School, State University of Campinas; Felipe T Galvão, PhD Student, Principal Investigator — Piracicaba Dental School, State University of Campinas; Thayane C Businari, PhD Student, Principal Investigator — Piracicaba Dental School, State University of Campinas; Raíssa Micaella M Machado, PhD, Principal Investigator — Piracicaba Dental School, State University of Campinas; Altair Antoninha D Cury, PhD, Principal Investigator — Piracicaba Dental School, State University of Campinas; Márcio Z Casati, PhD, Principal Investigator — Piracicaba Dental School, State University of Campinas
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No